CLINICAL TRIAL: NCT04380428
Title: Risk Literacy Among Portuguese Medical and Dentistry Students - a Cohort Study
Brief Title: Risk Literacy Among Portuguese Medical and Dentistry Students
Acronym: RiskommPt
Status: Completed | Type: Observational
Sponsor: Harding Center for Risk Literacy (Other)
Responsible Party: Principal Investigator, Niklas Keller, Principal Investigator, Harding Center for Risk Literacy
Other Study IDs: HC2019/11
Record Dates: First submitted 2020-05-04; First posted 2020-05-08 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Medical Education; Decision Support Techniques
Keywords: medical education; risk literacy; risk savvy; statistics; risk communication; probabilistic data; heuristics; students

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross section of the student body.: Matriculated students at Portuguese medical and dental faculties.
  Interventions: Other: No Intervention. Observational study.

INTERVENTIONS:
Other: No Intervention. Observational study. — No Intervention. Observational study.

SUMMARY:
This study is an online survey to assess risk literacy among students of the medical and dentistry faculties in Portugal. Risk literacy is the capability to understand and interpret statistical information, based on simple rules of thumb.

The investigators assess the level of "medical risk literacy" among Portuguese medical and dentistry students with the Quick Risk Test (QRT) and the multiple choice version of the Berlin Numeracy Test (BNT).

DETAILED DESCRIPTION:
This study is an online survey to assess risk literacy among students of the medical and dentistry faculties in Portugal.

The primary outcome is the measurement of "medical risk literacy" among Portuguese medical and dentistry students as assessed with the Quick Risk Test (QRT) and the multiple choice version of the Berlin Numeracy Test (BNT).

Secondary outcomes is to investigate whether study year, faculty, and prior statistical education have an impact on the level of risk literacy. Participants will be invited via email through established faculty mailing lists or established social media channels. For the survey, an online-survey tool (Unipark, academic program or Questback) will be used. Participation is voluntary and can be withdrawn at any time by aborting the survey (e.g. via closing the browser). Informed consent will be acquired at the beginning of the survey. English and Portuguese versions will be available to the participant.

As incentive to participate, participants completing the brief (ca.15 minutes) online-questionnaire will be granted a free subscriptions to the AMBOSS medical learning platform (2 weeks) and have the option to be entered into a lottery with the possibility of winning one of 3 free 6 month subscriptions.

After completion of the questionnaire, participants will be re-directed to a dedicated AMBOSS website where they can enter their email-address to take part in the lottery. This assures strict separation of the anonymous experimental data and the AMBOSS subscription data. Prior to initiation of the questionnaire, in the invitation email, participants will be provided the full participant information and made aware that, due to anonymity, it will not be possible to retrospectively delete their responses once the survey has been completed.

As the primary outcome is a baseline assessment and the secondary outcomes are exploratory analyses, no hypotheses will be tested in this survey.

ELIGIBILITY:
Inclusion Criteria:

* medical and dentistry students of Portuguese faculties
* active matriculation at a Portuguese faculty
* completion of the questionnaire

Exclusion Criteria:

* no active matriculation at a Portuguese faculty

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All matriculated students at Portuguese medical and dental faculties will be invited to participate (participation of faculties to be confirmed).
Sampling Method: Non-Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Quantitative measurement of "medical risk literacy" | 1st - 30st of May 2020
  Quantitative measurement of "medical risk literacy" among Portuguese medical and dentistry students measured with the Quick Risk Test (QRT) [Jenny, Keller & Gigerenzer, 2018] and the multiple choice version of the Berlin Numeracy Test (BNT) [Cokely & Galesic, 2012].

SECONDARY OUTCOMES:
Impact of study year, faculty, and prior statistical education on the level of risk literacy | 1st - 30st of May 2020
  Secondary outcomes is to investigate, whether study year, faculty, and prior statistical education have an impact on the level of risk literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Keller, Dr. rer. nat, Principal Investigator — Harding Center, Charité Universitätsmedizin Berlin, Germany; Alexej Zhogov, Principal Investigator — Harding Center for Risk Literacy, Charité Universitätsmedizin Berlin, Germany; Maxim Benz, Principal Investigator — Harding Center for Risk Literacy, Charité Universitätsmedizin Berlin, Germany; Mário Pereira Pinto, Dr., Principal Investigator — Presidency of the Portuguese Republic, Portugal; Henrique Proença da Cunha, Dr., Principal Investigator — Faculty of Medicine of the University of Coimbra, Portugal; Gerd Gigerenzer, Prof., Principal Investigator — Harding Center for Risk Literacy; Miriam Jenny, Dr., Principal Investigator — Harding Center for Risk Literacy
Locations (1):
- Harding Center for Risk Literacy, Potsdam, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
We plan to share our anonymized raw data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the completion of the study.
Access Criteria: undecided. Further research in risk literacy. For example other countries, or time delay. Or intervention studies.

REFERENCES:
- [Background] Jenny MA, Keller N, Gigerenzer G. Assessing minimal medical statistical literacy using the Quick Risk Test: a prospective observational study in Germany. BMJ Open. 2018 Aug 23;8(8):e020847. doi: 10.1136/bmjopen-2017-020847. PMID 30139896
- [Background] Correction: Assessing minimal medical statistical literacy using the Quick Risk Test: a prospective observational study in Germany. BMJ Open. 2018 Oct 18;8(10):e020847corr2. doi: 10.1136/bmjopen-2017-020847corr2. No abstract available. PMID 30341144
- [Background] Garcia-Retamero R, Cokely ET, Ghazal S, Joeris A. Measuring Graph Literacy without a Test: A Brief Subjective Assessment. Med Decis Making. 2016 Oct;36(7):854-67. doi: 10.1177/0272989X16655334. Epub 2016 Jun 27. PMID 27353824
- [Background] Lindskog M, Kerimi N, Winman A, Juslin P. A Swedish validation of the Berlin Numeracy Test. Scand J Psychol. 2015 Apr;56(2):132-9. doi: 10.1111/sjop.12189. Epub 2015 Jan 8. PMID 25581209
- [Background] Garcia-Retamero R, Galesic M, Gigerenzer G. Enhancing understanding and recall of quantitative information about medical risks: a cross-cultural comparison between Germany and Spain. Span J Psychol. 2011 May;14(1):218-26. doi: 10.5209/rev_sjop.2011.v14.n1.19. PMID 21568179
- [Background] Gigerenzer G, Wegwarth O. Five year survival rates can mislead. BMJ. 2013 Jan 29;346:f548. doi: 10.1136/bmj.f548. No abstract available. PMID 23360815
- [Background] Keller N, Feufel MA, Kendel F, Spies CD, Gigerenzer G. Training medical students how to extract, assess and communicate evidence from an article. Med Educ. 2017 Nov;51(11):1162-1163. doi: 10.1111/medu.13444. Epub 2017 Sep 7. No abstract available. PMID 28884483
- [Background] Wegwarth O, Wagner GG, Gigerenzer G. Can facts trump unconditional trust? Evidence-based information halves the influence of physicians' non-evidence-based cancer screening recommendations. PLoS One. 2017 Aug 23;12(8):e0183024. doi: 10.1371/journal.pone.0183024. eCollection 2017. PMID 28832633
- [Background] Caverly TJ, Prochazka AV, Combs BP, Lucas BP, Mueller SR, Kutner JS, Binswanger I, Fagerlin A, McCormick J, Pfister S, Matlock DD. Doctors and numbers: an assessment of the critical risk interpretation test. Med Decis Making. 2015 May;35(4):512-24. doi: 10.1177/0272989X14558423. Epub 2014 Nov 5. PMID 25378297
- [Background] Corrigendum: doctors and numbers: an assessment of the critical risk interpretation test. Med Decis Making. 2015 May;35(4):410. doi: 10.1177/0272989X15585799. No abstract available. PMID 25943577
- See also: Harding Center for Risk Literacy — https://www.hardingcenter.de/en

DOCUMENTS (1):
  • Study Protocol (2020-05-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT04380428/Prot_000.pdf